CLINICAL TRIAL: NCT06168825
Title: Mind Over Matter for Black and African American Women: A Single Arm Trial Examining Feasibility and Acceptability of a Supportive Intervention
Acronym: MOM
Status: Completed | Type: Observational
Sponsor: Inova Health Care Services (Other)
Collaborators: Howard University (Other); University of Louisville (Other); University of Houston (Other); VCU Massey Cancer Center (Unknown); Tigerlily Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: U23-06-5102
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Cancer; Breast Cancer; Brain Cancer; Central Nervous System Cancer; Colorectal Cancer; Esophageal Cancer; Gynecologic Cancer; Head and Neck Cancer; Gastrointestinal Cancer; Genitourinary Cancer; Melanoma; Blood Cancer; Lung Cancer; Acceptance and Commitment Therapy; Mind-Body Therapies; Psychosocial Intervention
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Brain Neoplasms; Central Nervous System Neoplasms; Colorectal Neoplasms; Esophageal Neoplasms; Head and Neck Neoplasms; Gastrointestinal Neoplasms; Urogenital Neoplasms; Melanoma; Hematologic Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Black and African American Women diagnosed with Cancer: Participants who have completed primary treatment (completed chemotherapy and/or radiation and/or surgery) are eligible to participate in the study
  Interventions: Other: Mind Over Matter (MOM)

INTERVENTIONS:
Other: Mind Over Matter (MOM) — Each participant's involvement in the study will include:
  * Attending a Pre-Program Orientation which will be held a week before the first MOM Session.
  * Completing 5 weekly sessions of MOM
  * Completing 2 surveys; one will be given before the start of the intervention (a pre-test) and the other will be given after the last MOM Session (a post-test)
  Participants will also have the option to participate in an optional Focus Group session which will occur a week after the last MOM Session ends
  Participants will spend about 6 weeks in this study. If they decide to participate in the optional session, they will spend about 7 weeks in this study.
  Please note, this entire Intervention will be offered online. There will be no in-person sessions or visits.

SUMMARY:
The goal of this study is to learn if the Mind Over Matter (MOM) Intervention, a 5-week group program, can help Black and African American women deal with the fears, worries and sadness that often accompany cancer diagnosis and treatment. The main question this study aims to answer is:

• Whether the MOM Intervention is feasible and acceptable among Black and African American women.

We would also like to find out if:

* The MOM Intervention decreases anxiety, depression and physical symptom severity for Black and African American women.
* The MOM Intervention is culturally and linguistically appropriate, and identify barriers, strengths, and areas of improvement.

Participants will:

* Attend a Pre-Program Orientation
* Attend 5 weekly MOM Sessions
* Complete 2 questionnaires (one will be given before the first MOM Session begins, and the other will be given after the last MOM Session)

Participants also have the choice to attend an optional Focus Group, which will be offered after the last MOM Session.

Please note, this entire Intervention will be offered online. There will be no in-person sessions or visits.

DETAILED DESCRIPTION:
Up to half of patients affected by cancer will experience psychosocial distress. Emotional and physical symptoms are two common facets of psychosocial distress. For those managing cancer, unmet psychosocial needs can lead to lower quality of life, poorer adherence to medical treatments, and increased healthcare costs. In a recent study investigating White, African American, Hispanic, Asian and Pacific Islander patients, it was found that African American patients were significantly more likely to experience clinical levels of psychosocial distress.

Inova Life with Cancer® has developed Mind Over Matter (MOM), a group psychosocial program designed to teach emotional coping skills to anyone affected by cancer. MOM consists of five, 1.5-hour sessions. The foundational theories of MOM are Cognitive Behavioral Therapy (CBT), Acceptance & Commitment Therapy (ACT), and the physiology of the stress response. Each session introduces a core cognitive concept and a different relaxation exercise. These sessions are structured and educational, with a focus on building skills, and are not a therapy or a support group. At the end of each session, participants are given exercises to practice the core cognitive concept and the relaxation at home. Participants are also offered optional reading to support the core cognitive concept. Practice outside of the class is vital. Thus, it is important to allow enough time to process and review the home practice exercises each week - this is the core of the program.

A retrospective secondary data analysis of the MOM intervention found a significant decrease in anxiety, depression, physical symptom severity, and physical symptom interference from pre- to post-test.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Black or African American
* Self-identify as female or a woman
* Having received a diagnosis and treatment for any type of cancer
* Having completed primary treatment (completed chemotherapy and/or radiation and/or surgery)
* ≥18 years of age
* Able to understand and provide valid informed consent prior to any study procedure
* Access to the internet and email
* Being able to speak and understand written and spoken English

Exclusion Criteria:

* Self-identify as other than Black or African American
* Does not Self-identify as a female or a woman
* Does not have a diagnosis of cancer
* Has not completed primary treatment
* Under the age of 18
* Not able to understand and provide valid informed consent
* Does not have access to the internet or email
* Not being able to speak, read and understand English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants who self-identify as female or a woman are eligible for the Intervention
Study Population: Patients will be recruited from the Howard University Cancer Center, a cancer center that treats patients that are primarily of African American descent in the Washington, DC metropolitan area, Inova Schar Cancer Institute, a state-of-the-art cancer center in the Washington, DC metropolitan area, and Inova Life With Cancer, a program of the Inova Schar Cancer Institute, which offers a variety of programs and services for cancer patients, survivors and their family members.
  The outreach for participants will be supported by collaborations and relationships with organizations and institutions that support Black and African American women managing cancer such as the Tigerlily Foundation and the VCU Massey Cancer Center.
  Potential Participants may also self-refer themselves to this study by contacting the study team.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Feasibility of MOM intervention | Baseline to 7 weeks
  The MOM intervention will be considered feasible if 60% of the participants registered to attend the intervention (and complete the consent process) complete 4 out of 5 sessions of the intervention
Acceptability of the MOM intervention | Baseline (pretest) and 7 weeks (posttest)
  Telehealth Usability Questionnaire (TUQ) which will be used to measure the primary endpoint of acceptability, the TUQ response set ranges from 1 (disagree) to 7 (agree). Anchoring the score of 4 as neither disagree or agree and 5, 6, and 7 are some levels of agreement. The MOM intervention will be considered acceptable if the average usability score, as measured by the TUQ, are equal to or above 4.5.

SECONDARY OUTCOMES:
Change in Depression from baseline | Baseline and 7 weeks
  Patient Health Questionnaire-8 (PHQ-8) self-report 9-item Likert scale will be used to measure Depression. The first eight items are scored from 0 (not at all) to 4 (nearly every day) with scores ranging from 0 to 32. The last item asks about how difficult the depression is in terms of daily functioning, using a scale from 0 (not at all) to 3 (extremely). The higher the score, the higher the depression. Change in Depression will be considered significant if the mean PHQ-8 scores decrease from the pre- to post-test.
Change in Anxiety from baseline | Baseline and 7 weeks
  The Generalized Anxiety Disorder 7 (GAD-7) will be used to measure anxiety. For the first 7 items scores range from 0 (not at all) to 3 (nearly every day) with scores ranges from 0 to 21. Item 8 asks how difficult anxiety has been in terms of daily functioning. The range of scores is 0-21, with the higher score being higher levels of anxiety being reported. Change in Anxiety will be considered significant if the mean GAD-7 scores decrease from the pre- to post-test.
Change in symptom severity from baseline | Baseline and 7 weeks
  The MD Anderson Symptom Inventory (MDASI) will be used to measure physical symptom severity and interference with daily living. The MDASI is made up of two subscales, the first includes 13 physical symptoms and the second includes six interference items. The physical symptom severity items are rated on an 11-point scale (0 = not present to 10 = as bad as you can imagine) and the interference items are rated on an 11-point scale (0 = did not interfere to 10 = interfered completely). For both subscales, the higher the score the worse the severity and the level of interference. Change in Symptom severity will be considered significant if the mean MDASI scores decrease from the pre- to post-test.
Number of participants who reported MOM intervention as Cultural appropriate | Baseline and 7 weeks
  Cultural appropriateness of the MOM intervention will be determined by participants' self-reported accounts
Number of participants who reported MOM intervention as linguistically appropriate | Baseline and 7 weeks
  linguistic appropriateness of the MOM intervention will be determined by participants' self-reported accounts

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Ferretti, MSW, LCSW, OSW-C, Principal Investigator — Inova Health Care Services
Locations (2):
- United States (2):
  - Howard University Cancer Center, Washington D.C., District of Columbia
  - Inova Life With Cancer, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ferretti M, Lowery Walker K, Bires J, BrintzenhofeSzoc K. Building coping skills to relieve distress and physical symptoms: Findings from a quality improvement project of a five-week group psychoeducational program for cancer patients. J Psychosoc Oncol. 2024;42(2):256-270. doi: 10.1080/07347332.2023.2238263. Epub 2023 Jul 24. PMID 37486181
- See also: Study Website — https://www.lifewithcancer.org/mind-over-matter-for-black-african-american-women/